CLINICAL TRIAL: NCT04620824
Title: TIssue Models for Invasive Disease (TIMID)
Acronym: TIMID
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Leicester (Other)
Collaborators: University Hospitals, Leicester (Other); University of Nottingham (Other)
Responsible Party: Sponsor
Other Study IDs: 0640
Record Dates: First submitted 2020-10-27; First posted 2020-11-09 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Spleen; Septic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Experiments include ex vivo organ perfusion and infection with bacteria or viruses. Biopsies of the perfused 24 spleens are processed for in vitro tissue slice and macrophage cell culture. The resulting primary cell cultures and tissue slices will be stored frozen for future research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Trial Participants: Overall Description of Trial Participants: The spleen organ samples included in this project will be from patients undergoing elective surgery for a lesion in the pancreas in the HPB Unit of the Leicester General Hospital. No change in the surgical procedure or recruiting results from this study and the use of the samples.
  Inclusion Criteria: The samples included in this project will be from patients undergoing elective surgery in the HPB Unit of the Leicester General Hospital. The criteria for inclusion of spleen samples from radical surgery are adult age and presence of splenic tissue in the discarded material after hepato-pancreato-biliary surgery.
  Exclusion Criteria: The main exclusion criterion is acute invasive bacterial and viral infection, but these patients are automatically excluded from major surgery. Vulnerable groups will not be recruited.

SUMMARY:
The human immune response to bacterial blood stream infection (sepsis) and systemic viral infection are fairly well understood, but we lack details on the most early phases. Better knowledge of these events would be important for the prevention and treatment of severe bacterial or viral disease. From models of infection, we have data showing that bacteria replicate in a specific type of cells in the spleen from where the bacteria then seed to the blood to cause blood stream infection. In order to gain more relevant data for humans, we have developed a spleen perfusion model using pig organs. This model confirms our previous work and most importantly will now allow us to study these events in human organs.

In order to move novel treatment strategies into human trials, we propose to test early events during infection using human spleens and the cells and tissues derived thereof. This research is expected to provide data on the relevance of the early events in bacterial and viral disease, in particular on the role of immune cells. The research includes work with human cells and tissue obtained from human spleens. In these settings, we will test pharmacological prevention and treatment of severe bacterial or viral infection (sepsis). The expected outcome of this work on human organs and tissue is expected to provide evidence that allows to move new treatment options into clinical trial.

This study is a preclinical research project and does not involve any intervention on patients, but it involves human tissue. The source of the human splenic tissue for our research will be spleen tissue removed during radical surgery. The present application relates exclusively to the ethical approval for the use of spleen tissue removed during radical surgery and discarded. The utilisation of the spleen or splenic tissue for research purposes does not alter in any way the surgical procedures at any stage and importantly the research will involve only anonymity samples.

DETAILED DESCRIPTION:
This is a preclinical research project and no patient intervention is planned. The project makes use of anonymised human tissue samples discarded during radical surgery. The spleen organ samples included in this project will be from patients undergoing elective surgery for a lesion in the pancreas in the HPB Unit of the Leicester General Hospital. The sample size of 100 (100 enrolled subjects for 42 spleens) has been determined by power calculations and is in line with the number of spleens actually removed by elective pancreas surgery over the past years. No change in the surgical procedure or recruiting results from this study and the use of the samples. All the experimental work carried out on the spleen samples will have no effect on the patient.

Experiments include ex vivo organ perfusion and infection with bacteria or viruses. Biopsies of the perfused 42 spleens are processed for in vitro tissue slice and macrophage cell culture. The resulting primary cell cultures and tissue slices will be stored frozen for future research. All in vitro studies on the 42 organs, and the tissues and cells derived from them, will evaluate the effect of therapeutic interventions (antibodies, receptor antagonists, antibiotics and other molecules) on the capacity of splenic cells to clear invasive bacteria or viruses. The experiments will be carried out each time a spleen sample will be available.

The detailed technical description of the experimental strategy including the strategy for storage and discarding of the human tissue will be as follows:

1. Whole organ ex vivo perfusion: This work is done to stabilise the organ, infect the organ and then to derive from it tissue slices and cells for primary cell culture. We have successfully set up a normo-thermic ex vivo porcine spleen perfusion model. This expertise allowed us to define the parameters for organ collection, transport and perfusion of porcine spleens for up to six hours and importantly develop and infection model. Infection showed conservation of capacity to remove bacteria from blood and good filtering capacity and, essential for this application, that also in the whole organ model specific subsets of macrophages are permissive to bacterial intracellular replication. In this experimental series we propose to perfuse whole explanted human spleens. In contrast to pigs, we will use for perfusion of the human organ synthetic medium in order to neutralise or minimise acquired immunity. Histology, confocal microscopy, FACS analysis aRNAseq of pathogens and host cells and bacterial, parasite and viral enumeration will be the main methodologies to analyse the perfused organ. The aim of this part of the work is to demonstrate that at the whole organ level bacteria and viruses are able to replicate in splenic tissue macrophages pinpointing attention of anti-infective treatments to the prevention of these early steps potentially preventing invasive bacterial and viral disease. Samples from the 42 whole perfused organs will be the source of tissue slice cultures and primary cell cultures.
2. Primary cell cultures: From the 42 human spleens we will derive samples for primary culture of human tissue macrophages and other immune cells. Using the methodology in use for cells from mice and pigs, we will set up primary cultures of human splenic immune cells and in particular macrophages. Immune cells including macrophages and neutrophils will be purified by different methodologies including by percoll gradient centrifugation, FACS and magnetic separation and cultured for up to seven days. Cultures will be tested for multiple parameters including cytokines, surface markers, anybody production and gene expression. To test interaction with bacteria or viruses, the cultured cells will be infected with a panel of bacterial and viral pathogens. Upon other methodology, confocal microscopy, FACS and RNAseq will be used monitor behaviour of bacterial, parasitic and viral pathogens and host cells. Interventions with cytokines, chemokines, drugs, antibiotics and other compounds will be carried out to test tractability of the system. With the aim in mind to identify targets for intervention, the cell culture models are intended to provide detailed quantifiable parameters of the interaction of bacteria or viruses and immune cells in particular tissue macrophages in a controlled in vitro culture system. This is intended to allow the design of medium-throughput assays to test strategies modifying initiation of invasive disease. Cells will be stored in liquid nitrogen for further research.
3. Organotypic slice cultures: From the 42 human spleens we will derive, in addition to cells, also tissue samples for organotypic slice cultures. With the methodology well set up for brain slices and described for spleen, we will culture organotypic human spleen slice cultures. These organ slices are superior to cell cultures, as they maintain the multicellular spatial microarchitecture of the organ, which is particularly important when analysing tissue macrophages. As for brain slice cultures, we will infect the slices with bacterial or viral pathogens and monitor their migration within the tissue, the infection of cells and the reaction of the single host cells. The use of tissue slice culture should allow to specifically study the targeting and replication-permissive nature of specific subsets of immune cells including macrophages. A goal of the objective is to allow for detailed development of infectious foci in the spleen including time laps confocal microscopy of infected spleen slices. Testing in this model cytokines and other host derived molecules are expected to show the potential of interventions targeting specific subsets of immune cells including macrophages. Tissue slices will be stored in liquid nitrogen for further research.

Sample transfer between units: The 42 planned organ perfusion will be performed at the laboratories of the HBP unit of the Leicester General Hospital. In selected cases organ perfusion might be performed at the Department of Genetics and Genome Biology of the University of Leicester. The relative HBA form has been obtained (Hazardous Biological Agents form GEN/45 Cell lines and primary human cell and tissue culture, date 02/10/2017). During and after perfusion, tissue samples for tissue slice culture and primary cell culture will be taken. These tissue samples will be transferred to the Department of Genetics and Genome Biology or Dept. of Infection and Immunity and Inflammation for the scheduled research work and will be stored there in accordance with regulations relative to the Human Tissue Act. Stored tissue slices and primary cell cultures may then be transferred for immunological studies to the University of Nottingham for experimental work detailed above for cell cultures. Conditions for handling, storage and transport are defined by the HBA form GEN45 and transfer will be regulated by an MTA.

ELIGIBILITY:
Inclusion Criteria:

* The samples included in this project will be from patients undergoing elective surgery in the HPB Unit of the Leicester General Hospital.
* Spleen samples from radical surgery are adult age (18-80 years)
* Presence of splenic tissue in the discarded material after hepato-pancreato-biliary surgery.

Exclusion Criteria:

* The main exclusion criterion is acute invasive bacterial and viral infection, but these patients are automatically excluded from major surgery.
* Samples from patients treated with antibiotics prior to explant or surgery will not be excluded, but samples will have to be tested for residual antibiotic activity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The spleen organ samples included in this project will be from patients undergoing elective surgery for a lesion in the pancreas in the HPB Unit of the Leicester General Hospital. No change in the surgical procedure or recruiting results from this study and the use of the samples.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2018-08-03 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary Objective | 3.5 Years
  The primary objective of the study is to identify therapies acting on the initial events during invasive bacterial and viral infection.

SECONDARY OUTCOMES:
Secondary Objectives | 3.5 Years
  The secondary objective of this study is to provide novel in vitro and ex vivo models of human splenic macrophages to study the impact of therapies for invasive infection.

CONTACTS AND LOCATIONS:
Locations (1):
- UHL NHS Trust - Leicester General Hospital, Leicester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Carreno D, Wanford JJ, Jasiunaite Z, Hames RG, Chung WY, Dennison AR, Straatman K, Martinez-Pomares L, Pareek M, Orihuela CJ, Restrepo MI, Lim WS, Andrew PW, Moxon ER, Oggioni MR. Splenic macrophages as the source of bacteraemia during pneumococcal pneumonia. EBioMedicine. 2021 Oct;72:103601. doi: 10.1016/j.ebiom.2021.103601. Epub 2021 Oct 4. PMID 34619637